CLINICAL TRIAL: NCT00393029
Title: Phase II Study of Metastatic Cancer That Overexpresses p53 Using Lymphodepleting Conditioning Followed by Infusion of Anti-p53 T Cell Receptor (TCR)-Gene Engineered Lymphocytes
Brief Title: Phase II Study of Metastatic Cancer That Overexpresses P53 Using Lymphodepleting Conditioning Followed by Infusion of Anti-P53 TCR-Gene Engineered Lymphocytes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Steven A. Rosenberg, M.D., Ph.D., National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 070003; 070003 (Other: National Institutes of Health (NIH)); 07-C-0003 (Other: National Institutes of Health (NIH))
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Results first posted 2011-08-05 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2011-08

CONDITIONS: Anti-p53 TCR-Gene
Keywords: Tumor Regression; In Vivo Cell Survival; Toxicity Profile; Metastatic Renal Cell Cancer; Cancer; Metastatic Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms; Neoplasm Metastasis | interventions — Genes, p53; tumor protein 53-induced nuclear protein 1, mouse; aldesleukin; Interleukin-2; Filgrastim; Granulocyte Colony-Stimulating Factor; Cyclophosphamide; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with metastatic melanoma (Experimental): Melanoma is a serious form of skin cancer that develops in the skin cells that make our skin color (melanocytes).
  Interventions: Biological: anti-protein 53 or tumor protein 53 (p53) T-cell receptor transduced peripheral blood lymphocytes; Biological: aldesleukin; Biological: filgrastim; Drug: cyclophosphamide; Drug: fludarabine phosphate
- Patients with other metastatic cancers (Experimental)
  Interventions: Biological: anti-protein 53 or tumor protein 53 (p53) T-cell receptor transduced peripheral blood lymphocytes; Biological: aldesleukin; Biological: filgrastim; Drug: cyclophosphamide; Drug: fludarabine phosphate

INTERVENTIONS:
Biological: anti-protein 53 or tumor protein 53 (p53) T-cell receptor transduced peripheral blood lymphocytes — Peripheral blood lymphocytes are harvested by lymphapheresis and engineered to express a T cell receptor that binds to P53.
  Other Names: Tumor protein 53; Anti-protein 53
Biological: aldesleukin — 720,000 IU/kg intravenously over 15 minutes every 8 hours for up to 5 days
  Other Names: Interleukin-2 (IL-2); Proleukin; Recombinant human interleukin-2
Biological: filgrastim — Beginning on day 1 or 2, administered subcutaneously at a dose of 5 mcg/kg/day (not to exceed 300 mcg/day); continue daily until neutrophil count > 1.0 x 10^9/L x 3 days or > 5.0 x 10^9/L.
  Other Names: Granulocyte colony stimulating factor (GCSF); Neupogen
Drug: cyclophosphamide — 60 mg/kg/day x 2 days intravenously in 250ml dextrose 5% in water (D5W) with mesna 15 mg/kg/day x 2 days over 1 hour.
  Other Names: Cytoxan; Endoxan; Neosar; Procytox; Revimmune
Drug: fludarabine phosphate — 25 mg/m2/day intravenously piggyback (IVPB) daily over 30 minutes for 5 days.
  Other Names: Fludara

SUMMARY:
Background:

The p53 gene normally suppresses tumor growth, but when it is mutated, or damaged, tumors can grow unchecked.

In cancers where the p53 gene has mutated, an increased level of p53(overexpression of p53) can be measured in the tumor.

Objectives To determine whether advanced cancers that overexpress p53 can be treated effectively with lymphocytes (white blood cells) that have been genetically engineered to contain an anti-p53 protein.

Eligibility Patients 18 years of age and older with metastatic cancer (cancer that has spread beyond the original site) Patient's tumor overexpresses p53 Patient's leukocyte antigen type is HLA-A 0201 Design

Patients undergo the following procedures:

Leukapheresis (on two occasions). This is a method of collecting large numbers of white blood cells. The cells obtained in the first leukapheresis procedure are grown in the laboratory, and the anti-p53 protein is inserted into the cells using an inactivated (harmless)virus in a process called transduction. Cells collected in the second leukapheresis procedure are used to evaluate the effectiveness of the study treatment.

Chemotherapy. Patients are given chemotherapy through a vein (intravenously, IV) for 1 week to suppress the immune system so that the patients immune cells do not interfere with the treatment.

Treatment with anti-p53 cells. Patients receive an IV infusion of the transduced cells containing anti-p53 protein, followed by infusions of a drug called IL-2, which helps boost the effectiveness of the transduced white cells.

Patients may undergo a tumor biopsy (removal of a small piece of tumor tissue). Patients are evaluated with laboratory tests and imaging tests, such as computed tomography (CT) scans 4 to 6 weeks after treatment and then once a month 3 to 4 months to determine the response to treatment.

Patients have blood tests at 1, 3, 6 and 12 months and then annually for the next 10 years.

DETAILED DESCRIPTION:
Background:

Human peripheral blood lymphocytes (PBL's) can be engineered to express alpha T-cell receptor that recognizes an human leukocyte antigen serotype witin HLA-A A serotype group) HLA-A2. 1 restricted epitope derived from the p53 protein.

We constructed a single retroviral vector that contains both alpha and existent chains and can mediate genetic transfer of this TCR with high efficacy (less than 30%) without the need to perform any selection.

In co-cultures with HLA-A2 and p53 double positive tumors including melanoma, hepatoma, sarcoma, small-cell lung cancer, esophageal and breast tumors, p53-TCR transduced T cells secreted significant amount of IFN-(but no significant secretion was observed in control co-cultures with either HLA-A2+/p53- or HLA-A2-p53+cell lines.

Additional secretion of cytokines (IL-2, IL-4, IL-10,granulocyte macrophage stimulating factor (GM-CSF),tumor necrosis factor alpha (TNFalpha)) and chemokines (regulated upon activation, normal T cell expressed and secreted (RANTES), macrophage inflammatory protein 1 alpha (MIP-1 alpha)) was also observed in co-cultures with HLA-A2+/p53+tumor lines.

p53-TCR transduced PBL could efficiently kill HLA-A2, 1/p53 expressing tumors (H2087, MDA-MB 231, Saos2/143, BE-3).

In addition, we also tested for specific lysis of normal tissues by p53-TCR transduced cells and there was little or no lysis of the normal fibroblasts, renal epithelia cells, resting or activated normal PBLs compared to control HLA_A2+/p53+H2087 tumor.

Objectives:

Primary objective:

Determine of the administration of anti-p53 TCR-engineered peripheral blood lymphocytes and aldesleukin to patients following a nonmyeloablative but lymphoid depleting preparative regimen will result in clinical tumor regression in patients with metastatic cancer overexpressing p53.

Secondary objectives:

Determine the in vivo survival of TCR gene-engineered cells. Determine the toxicity profile of this treatment regimen.

Eligibility:

Patients who are HLA A0201 and 18 years of age or older must have metastatic cancer whose tumors overexpress p53; previously received and have been a non-responder or recurred to standard care for metastatic disease; biopsy available to evaluate p53 expression; normal values for basic laboratory values; Patients may not have: concurrent major medical illnesses; any form of primary or secondary immunodeficiency; severe hypersensitivity to any of the agents used in this study; contraindications for high dose aldesleukin administration.

Design:

PBMC, obtained by leukapheresis (approximately 5 x 10^9 cells) will be cultured in the presence of anti-CD3 Muromonab-CD3( OKT3) and IL-2 in order to stimulate T-cell growth.

Transduction is initiated by exposure of approximately 10^8 to 5 x 10^8 cells to supernatant containing the anti-p53 TCR retroviral vector. These transduced cells will be expanded and tested for their anti-tumor activity.

Patients will receive a nonmyeloablative but lymphocyte depleting preparative regiment consisting of cyclophosphamide and fludarabine followed by intravenous infusion of in vitro tumor reactive, TCR gene-transduced PBL plus IV aldesleukin (720,000IU/kg q8h for a maximum of 15 doses).

Patients will undergo complete evaluation of tumor with physical examination, CT of the chest, abdomen and pelvis and clinical laboratory evaluation four to six weeks after treatment and then monthly for approximately 3 to 4 months or until off study criteria are met.

Patients will be entered into two cohorts based on histology: cohort 1 will include patients with metastatic melanoma or renal cell cancer, cohort 2 will include patients with other types of metastatic cancer.

For each of the 2 strata evaluated, the study will be conducted using a phase II optimal design where initially 21 evaluable patients will be enrolled. For each of these two arms of the trial, if 0 or 1 of the 21 patients experiences a clinical response, then no further patients will be enrolled but if 2 or more of the first 21 evaluable patients enrolled have a clinical response, then accrual will continue until a total of 41 evaluable patients have been enrolled in that stratum.

For both strata, the objective will be to determine if the combination of high dose aldesleukin, lymphocyte depleting chemotherapy, and anti-p53 TCR-gene engineered lymphocytes is able to be associated with a clinical response rate that can rule out 5% (p0=0.05) in favor of a modest 20% PR + CR rate (p1=0.20).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have metastatic cancer that overexpresses p53 as assessed by immunohistochemistry, as determined by positive staining of tumor sample. when compared to negative controls per procedure in Appendix 1. The immunohistochemical staining will be performed in the Pathology Laboratory Center for Cancer Research (CCR), National Cancer Institute (NCI) on fresh or archival tissue and will be supervised by Dr. Maria Merino. The criteria used to determine overexpression will be that used in the Laboratory of Dr. Curt Harris. Ten fields will be evaluated at 40 X magnification and if greater than 5% of cells stain positive, the tumor will be categorized as an overexpressor.
* Patients with melanoma or renal cell cancer must have previously received interleukin-2 (IL-2) and have been either non-responders (progressive disease) or have recurred. Patients with other histologies,not including hematologic malignancies, must have previously received first line and second line or higher systemic standard care(or effective salvage chemotherapy regimens) for metastatic disease,if known to be effective for that disease and have been either non-responders (progressive disease) or have recurred.
* Age greater than or equal to 18 years.
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 to 1.
* Life expectancy of greater than three months.
* Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune competence and thus be less responsive to the experimental and more susceptible to its toxicities).
* Seronegative for hepatitis B antigen and hepatitis C antibody unless antigen negative.
* Patients must be human leukocyte antigen A(HLA-A) 0201 positive.
* Patients of both genders must be willing to practice birth control for four months after receiving the preparative regimen.
* Absolute neutrophil count greater than 1000/mm^3, and normal white blood cells (WBC) (greater than 3000/mm^3).
* Platelet count greater than 100,000/mm^3.
* Hemoglobin greater than 8.0 g/dl.
* Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than the upper limit of normal.
* Serum creatinine less than or equal to 1.6 mg/dl.
* Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
* More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo). Six weeks must have elapsed since prior Ipilimumab (MDX-010) therapy to allow antibody levels to decline, and patients who have previously received MDX-010 must have a normal colonoscopy with normal colonic biopsies.
* Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the preparative chemotherapy on the fetus.
* A biopsy must be evaluable to evaluate p53 expression and to confirm the diagnosis by the Laboratory of Pathology, CCR, NCI.

Exclusion Criteria:

* Patients requiring systemic steroid therapy
* Patients with active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
* Patients with any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease and acquired immune deficiency syndrome (AIDS)). Patients with opportunistic infections will be excluded. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
* Patients with history of severe immediate hypersensitivity reaction to any of the agents used in this study.
* Patient is not willing to sign a durable power of attorney.
* Patient is not able to understand and sign the Informed Consent Document.
* Since aldesleukin will be excluded if they have a history of electrocardio- gram (EKG) abnormalities, symptoms of cardiac ischemia or arrhythmias and have a left ventricular ejection fraction (LVEF) less than 45% on a cardiac stress test (stress thallium, stress multi-gated acquisition scan (MUGA), dobutamine echocardiogram, or other stress test).
* Similarly, patients who are greater than or equal to 50 years old with a LVEF less than 45% will be excluded.
* Patients with a prolonged history of cigarette smoking (greater than 20 pack/year within the past 2 years) or symptoms of respiratory dysfunction (e.g. grade 2 dyspnea or hypoxia) who do not have a normal pulmonary function test as evidenced by a FEV(1) less than 60% predicted will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Ph.D, Principal Investigator — NCI, NIH
Locations (1):
- National Institutes of Health, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kawakami Y, Eliyahu S, Delgado CH, Robbins PF, Rivoltini L, Topalian SL, Miki T, Rosenberg SA. Cloning of the gene coding for a shared human melanoma antigen recognized by autologous T cells infiltrating into tumor. Proc Natl Acad Sci U S A. 1994 Apr 26;91(9):3515-9. doi: 10.1073/pnas.91.9.3515. PMID 8170938
- [Background] Kawakami Y, Eliyahu S, Sakaguchi K, Robbins PF, Rivoltini L, Yannelli JR, Appella E, Rosenberg SA. Identification of the immunodominant peptides of the MART-1 human melanoma antigen recognized by the majority of HLA-A2-restricted tumor infiltrating lymphocytes. J Exp Med. 1994 Jul 1;180(1):347-52. doi: 10.1084/jem.180.1.347. PMID 7516411
- [Background] Kawakami Y, Eliyahu S, Delgado CH, Robbins PF, Sakaguchi K, Appella E, Yannelli JR, Adema GJ, Miki T, Rosenberg SA. Identification of a human melanoma antigen recognized by tumor-infiltrating lymphocytes associated with in vivo tumor rejection. Proc Natl Acad Sci U S A. 1994 Jul 5;91(14):6458-62. doi: 10.1073/pnas.91.14.6458. PMID 8022805
- See also: Medline Plus — http://www.nlm.nih.gov/medlineplus/
- See also: Drug Information — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: Genetics Home Page — http://ghr.nlm.nih.gov/
- See also: U S FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks
- See also: RECIST criteria — http://ctep.cancer.gov/protocolDevelopment/default.htm#protocol_development

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Expect to enroll 4-5 patients of each allowed histology up to a total of 82 patients. Approximately two years may be needed to accrue the maximum number of required patients.
Groups:
- Metastatic Melanoma: Melanoma is a serious form of skin cancer that develops in the skin cells that make our skin color (melanocytes).
Period: Overall Study
Arm/Group | Metastatic Melanoma | Other Metastatic Cancers
Started | 2 | 10
Completed | 2 | 9
Not Completed | 0 | 1
Not completed — Not treated | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metastatic Melanoma | Other Metastatic Cancers | Total
Number analyzed (Participants) | 2 | 10 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 10 | 12
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 44.5 (16.3) | 45.4 (9.2) | 44.95 (12.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 7 | 7
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 10 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 10 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 10 | 12

OUTCOME MEASURES:

1. Primary Outcome: Clinical Tumor Regression
Description: Response Evaluation Criteria In Solid Tumors (RECIST).
  See the protocol Link module for full criteria if desired.
Time Frame: 1-11 months
Measure: Number; unit: Participants
Groups:
- Metastatic Melanoma & Other Metastatic Cancers: Melanoma is a serious form of skin cancer that develops in the skin cells that make our skin color (melanocytes).
  There are no statistical differences between the arms, therefore, they can be combined for this outcome measure.
Arm/Group | Metastatic Melanoma & Other Metastatic Cancers
Number analyzed (Participants) | 9
Participants | 1

2. Primary Outcome: The Number of Participants With Adverse Events
Description: Here are the total number of participants with adverse events. Adverse events were described using the Common Terminology Criteria for Adverse Events (CTCAE) version 3. For the detailed list of adverse events see the adverse event module.
Time Frame: events related to all components of the treatment regimen were reported from the start of the non-myeloablative conditioning regiment through 30 days following treatment or resolution.
Measure: Number; unit: participants
Arm/Group | Metastatic Melanoma | Other Metastatic Cancers
Number analyzed (Participants) | 2 | 9
participants | 2 | 9

3. Secondary Outcome: In Vivo Survival of T-cell Receptor (TCR) Gene-engineered Cells in Participants
Description: Survival of TCR gene-engineered cells is defined as >10% murine TCR positive cells.
Time Frame: 3-12 months
Measure: Number; unit: participants
Arm/Group | Metastatic Melanoma | Other Metastatic Cancers
Number analyzed (Participants) | 2 | 9
participants | 2 | 9

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Metastatic Melanoma | Other Metastatic Cancers
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/9
Other Adverse Events (participants affected / at risk) | 2/2 | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metastatic Melanoma (N=2) | Other Metastatic Cancers (N=9)
BLOOD/BONE MARROW-Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 7 (9)
BLOOD/BONE MARROW - Leukocyte count decreased (Blood and lymphatic system disorders) | 2 (2) | 9 (13)
BLOOD/BONE MARROW-Lymphocyte count decreased (Blood and lymphatic system disorders) | 2 (2) | 9 (15)
BLOOD/BONE MARROW-Neutrophil count decreased (Blood and lymphatic system disorders) | 2 (2) | 9 (11)
BLOOD/BONE MARROW -Platelet count decreased (Blood and lymphatic system disorders) | 2 (2) | 9 (10)
CARDIAC GENERAL - Hypotension (Cardiac disorders) | 1 (1) | 1 (1)
COAGULATION - Activated partial thromboplastin time prolonged (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
CONSTITUTIONAL SYMPTOMS- Fatigue (General disorders) | 1 (1) | 4 (4)
CONSTITUTIONAL SYMPTOMS - Fever (General disorders) | 1 (1) | 4 (5)
DERMATOLOGY/SKIN-Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
GASTROINTESTINAL - Nausea (Gastrointestinal disorders) | 2 (2) | 6 (8)
GASTROINTESTINAL - Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (5)
HEMORRHAGE/BLEEDING - Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HEMORRHAGE/BLEEDING-Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
METABOLIC/LABORATORY-Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
METABOLIC/LABORATORY - Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
METABOLIC/LABORATORY-Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1) | 2 (4)
METABOLIC/LABORATORY - Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
METABOLIC/LABORATORY - Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (3)
NEUROLOGY - Confusion (Psychiatric disorders) | 1 (1) | 3 (3)
PAIN - Headache (Nervous system disorders) | 1 (1) | 6 (7)
VASCULAR-Capillary leak syndrome (Vascular disorders) | 1 (1) | 4 (5)
CARDIAC ARRHYTHMIA - Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
CONSTITUTIONAL SYMPTOMS-General symptom (General disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL- Anorexia (Gastrointestinal disorders) | 0 (0) | 2 (2)
GASTROINTESTINAL-Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL- Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL - Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
HEMORRHAGE/BLEEDING- Petechiae (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
INFECTION - Febrile neutropenia (Infections and infestations) | 0 (0) | 3 (3)
INFECTION- Sepsis (Infections and infestations) | 0 (0) | 1 (1)
INFECTION -Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
NEUROLOGY -Mini mental status examination abnormal (Nervous system disorders) | 0 (0) | 2 (3)
NEUROLOGY- Anxiety (Nervous system disorders) | 0 (0) | 1 (1)
PAIN - Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
PAIN - Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
PAIN - Breast pain (Reproductive system and breast disorders) | 0 (0) | 2 (2)
PAIN- Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN-Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN -Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
PAIN - Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
PAIN-Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PULMONARY/UPPER RESPIRATORY - Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY/UPPER RESPIRATORY- Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SECONDARY MALIGNANCY - Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No